CLINICAL TRIAL: NCT03541135
Title: Study on Cardiovascular Health, Nutrition and Physical Functioning in Older Adults in Spain (Seniors-ENRICA II)
Brief Title: Study on Cardiovascular Health, Nutrition and Physical Functioning in Older Adults in Spain
Acronym: Sen-ENRICAII
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Fernando Rodríguez-Artalejo, Professor of Preventive Medicine and Public Health, Universidad Autonoma de Madrid
Other Study IDs: Seniors-ENRICA II
Record Dates: First submitted 2018-03-20; First posted 2018-05-30 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Physical Disability; Cognitive Dysfunction
Keywords: Cardiovascular health; Diet; Functional limitations; Frailty; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Population aging makes it necessary to identify factors related to unhealthy aging. The purpose of this study is to examine the association between ideal cardiovascular health, diet and other lifestyles and biological risk factors (either clasical or emergent) and the risk of physical and cognitive function impairment and mortality in a cohort of community-living individuals aged 65 years and over.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized residents in the region of Madrid, Spain.
* 65 years and over

Exclusion Criteria:

* None

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-living individuals in the region of Madrid, Spain, aged 65 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Functional limitations on bicep-femoral flexibility | 3 years
  Chair Sit and Reach test
Functional limitations on shoulder flexibility | 3 years
  Back Scratch test
Functional limitations on balance | 3 years
  Short Physical Performance Battery (SPPB): Balance test
Functional limitations on gait speed | 3 years
  Short Physical Performance Battery (SPPB): Gait Speed test
Functional limitations on strength of legs | 3 years
  Short Physical Performance Battery (SPPB): Chair Stand test
Functional limitations on strength of hands | 3 years
  Hydraulic hand dynamometer (Jamar Plus +)
Functional limitations on activities of daily living | 3 years
  Activities of Daily Living (ADLs) test
Functional limitations on instrumental activities of daily living | 3 years
  Instrumental Activities of Daily Living (IADLs) test
Functional limitations on olfactory function | 3 years
  Pocket Smell test
Functional limitations on taste function | 3 years
  NIH Tool Box Taste test
Functional limitations on auditory function | 3 years
  Audiometry
Cognitive impairment | 3 years
  Mini-Mental State Examination (MMSE)
Executive function limitations on working memory | 3 years
  Digits Forward test (WAIS-III),
Executive function limitations on programmed motor tasks | 3 years
  Three Hand Position test of Luria
Executive function limitations on motor response control | 3 years
  GO-NO-GO test.
Memory function limitations | 3 years
  Seven Minute Screen (orientation, memory, clock drawing, verbal fluency)
Frailty | 3 years
  Fried criteria
Falls | 3 years
  From the question:
  "How many times have you fallen down since the last interview? a) Number of falls; b) Number of injurious falls; c) Number of falls with fracture
Arterial stiffness estimated by pulse wave velocity (PWV) | 3 years
  Ambulatory Blood Pressure Monitor using the oscillometric method (Mobil-O-Graph PWA) to estimate PWV (m/s) over a 24 hours period
Arterial stiffness estimated by central sistolic blood pressure (CSBP) | 3 years
  Ambulatory Blood Pressure Monitor using the oscillometric method (Mobil-O-Graph PWA) to estimate CSBP (mmHg) over a 24 hours period
Arterial stiffness estimated by augmentation index (AI) | 3 years
  Ambulatory Blood Pressure Monitor using the oscillometric method (Mobil-O-Graph PWA) to estimate AI (%) over a 24 hours period
24-h systolic and diastolic blood pressure | 3 years
  Ambulatory Blood Pressure Monitor using the oscillometric method (Mobil-O-Graph PWA) to estimate brachial blood pressure (systolic and diastolic) (mmHg) over a 24 hours period
Mortality | 3 years
  From the National Institute of Statistics of Spain

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rodríguez-Artalejo, MD, PhD, Principal Investigator — Department of Preventive Medicine and Public Health. Universidad Autónoma de Madrid; Jose R Banegas, MD, PhD, Principal Investigator — Department of Preventive Medicine and Public Health. Universidad Autónoma de Madrid
Locations (1):
- Department of Preventive Medicine and Public Health. Universidad Autonoma de Madrid, Madrid, Spain

REFERENCES:
- [Derived] Marcos-Delgado A, Yevenes-Briones H, Fernandez-Villa T, Martin-Sanchez V, Guallar-Castillon P, Rodriguez-Artalejo F, Lopez-Garcia E. Association between diet quality and malnutrition: pooled results from two population-based studies in older adults. BMC Geriatr. 2024 May 10;24(1):417. doi: 10.1186/s12877-024-04984-5. PMID 38730363
- [Derived] Vega-Cabello V, Struijk EA, Caballero FF, Lana A, Arias-Fernandez L, Banegas JR, Rodriguez-Artalejo F, Lopez-Garcia E. Dietary Micronutrient Adequacy and Risk of Multimorbidity in Community-dwelling Older Adults. Am J Clin Nutr. 2023 Jul;118(1):34-40. doi: 10.1016/j.ajcnut.2023.05.008. Epub 2023 May 3. PMID 37146761